CLINICAL TRIAL: NCT03414385
Title: Epigenomic Remodeling of Metabolism by Exercise
Brief Title: Effect of Exercise on Genes That Control Muscle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dennis T. Villareal, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-40366; 1R01DK111436-01A1 (NIH)
Record Dates: First submitted 2018-01-17; First posted 2018-01-29 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): Research volunteers will be asked to undergo an acute bout of aerobic exercise at moderate intensity for ~120 minutes. Before and after the exercise the volunteer will undergo leg biopsy.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Acute bout of aerobic exercise at moderate intensity for 2 hours

SUMMARY:
The proposed project will examine how exercise counteracts metabolic disorders and type 2 diabetes through regulating gene expression. The project is highly relevant to public health because of the global pandemic of diabetes, obesity, and associated metabolic syndromes as well as the well-known metabolic benefit of physical exercise in correcting these disorders.

DETAILED DESCRIPTION:
Exercise is a first-line treatment for type 2 diabetes, and exerts its beneficial effects not only by burning off energy but also by causing prolonged metabolic changes through changing gene expression. Genes are our genetic materials and the expression of genes determines our biology. In our previous study in animals, we identified some factors that drive exercise-induced gene expression changes. Here we would like to address whether the result is also true in human. This work will provide molecular insights into how exercise remodels our metabolism and will potentially find a way to maximize the benefit we get from physical exercise.

The purpose of this study is to determine whether acute exercise activate certain molecular factors in human skeletal muscle. Participants will be asked to undergo an acute bout of aerobic exercise at ~ moderate intensity for about 2 hours. Before and after the exercise, the participants will undergo a muscle biopsy. The muscle tissues will be used for total RNA extraction and RT-qPCR analysis of genes that include but are not limited to de facto JunD/AP-1 target genes and will also be analyzed by Jun D Chip-qPCT to assess binding of Jun D on its de facto target genes.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 40 years
* BMI 18.5 - 29.9
* Stable body weight (not more than 2 kg change) during the past 6 months
* Moderate sedentary (regular exercise less than 1 hour per week for the last 6 months)
* Willing to provide informed consent

Exclusion Criteria:

* Failure to provide informed consent
* Any major chronic disease or any condition that would interfere with exercise, in which exercise is contraindicated, or that would interfere with interpretation of results
* Severe orthopedic and or neuromuscular disease that would contraindicate participation in exercise
* Other significant co-morbid disease that would impair ability to exercise
* Uncontrolled hypertension (BP greater than 160/90)
* History of malignancy during the past 5 years
* Diabetes mellitus as determined by self-report with verification (medical records, current treatment, confirmation from health care provider), or HbA1c of exceeding 6.5%

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in JunD/AP-1 signaling in human skeletal muscle | Immediately after about 2 hours exercise
  JunD/AP-target genes

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD, Principal Investigator — Baylor College of Medicine; Zheng Sun, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine/Michael E DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No